CLINICAL TRIAL: NCT02744586
Title: A Randomized Control Study to Evaluate Novel Interventions to Reduce Risk Factors Associated With HIV, Neglected Tropical and Non-communicable Diseases Among Couples in Zambia
Brief Title: Zambia One Love Aim 3 Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Susan Allen, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00083001
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: HIV; Sexually Transmitted Diseases; Neglected Diseases; Non-communicable Diseases
Keywords: Sexually transmitted infections; Neglected tropical diseases; Non-communicable diseases
MeSH Terms: conditions — Sexually Transmitted Diseases; Neglected Diseases; Noncommunicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strengthening our Vows (SOV) Group (Experimental): Participants in the SOV arm will participate in the "Together HIV Free" and "Protecting My Spouse" plans.
  Interventions: Behavioral: Strengthening Our Vows (SOV)
- Good Health Package Plus (GHPP) Group (Placebo Comparator): Participants in the GHPP arm will receive education on the prevention of helminths, schistosomiasis, hypertension, diabetes, and diarrheal diseases through participatory and interactive group sessions.
  Interventions: Behavioral: Good Health Package Plus (GHPP)

INTERVENTIONS:
Behavioral: Strengthening Our Vows (SOV) — Participants, led by a counselor, will discuss options to keep HIV from entering their relationship including both sex partners remaining monogamous, using condoms every time they have sex with outside partners, and being tested together with outside partners to ensure they are HIV negative (Together HIV Free Plan). Participants will discuss options in the event of an outside exposure to HIV including abstaining from having sex with their spouse or by using condoms every time they have sex with their spouse until they can be retested for HIV after 30 days (Protecting my Spouse Plan).
  Participants will be screened for hypertension, diabetes, schistosomiasis, HIV, syphilis, and trichomonas vaginalis and the presence of sperm (women only). Health problems will be treated or referred. Couples will be administered questionnaires that record self-report of sexually transmitted infections, number of outside partners, and reports of sex without a condom with outside partners.
  Arms: Strengthening our Vows (SOV) Group
Behavioral: Good Health Package Plus (GHPP) — Participants, led by a counselor, will discuss how to prevent, screen, and treat neglected tropical diseases (helminths and schistosomiasis), non-communicable diseases (hypertension and diabetes) and diarrheal diseases through basic hygiene and sanitation. The facilitator will demonstrate proper handwashing techniques and chlorination of water and discuss diet and lifestyle changes. Participants will be screened for hypertension, diabetes, schistosomiasis, HIV, syphilis, and trichomonas vaginalis and the presence of sperm (women only). Health problems will be treated or referred. Couples will also be administered questionnaires that record self-report of sexually transmitted infections, number of outside partners, and reports of sex without a condom with outside partners.
  Arms: Good Health Package Plus (GHPP) Group

SUMMARY:
The aim of this study is to determine whether a Strengthening our Vows (SOV) intervention will reduce HIV exposures from concurrent partnership (CP) when compared to the control Good Health Package Plus (GHPP), in addition to couples' voluntary HIV counseling and testing (CVCT), among concordant HIV-negative couples living in Zambia.

DETAILED DESCRIPTION:
This is a randomized control study to evaluate novel interventions to reduce risk factors associated with HIV, neglected tropical and non-communicable diseases among couples in Zambia.

The aim of this study is to determine whether a Strengthening our Vows (SOV) intervention will reduce HIV exposures from concurrent partnership (CP) when compared to the control Good Health Package Plus (GHPP), in addition to couples' voluntary HIV counseling and testing (CVCT), among concordant HIV-negative couples.

Investigators seeks to compare the impact of the SOV intervention and the GHPP intervention on reduction in a composite of risk factors associated with HIV acquisition from concurrent partners, compare the impact of GHPP and SOV on knowledge and use of hygiene and sanitation measures and hypertension and diabetes screening and management, and compare self-reported couples' testing (CVCT) with outside partners in the SOV and GHPP arms.

Couples will receive SOV or GHPP based on the pre-randomization of the clinic which they attend for standard of care HIV counseling and testing. The Strengthening our Vows (SOV) intervention will seek to establish a dialogue or norm where couples will be able to protect each other from HIV infection from outside partners. The Good Health Package Plus (GHPP) intervention focuses on strategies to improve household health related to diarrheal diseases, helminths, schistosomiasis, diabetes, and hypertension.

ELIGIBILITY:
Inclusion Criteria:

Heterosexual Zambian couples who have undergone CVCT as standard of care in government health clinics in Lusaka and Ndola. Couples must be women 18-45 cohabiting with men 18-65 years old, have cohabited 3 months or greater, are both HIV-negative and are able to attend the scheduled follow-up visits.

* Heterosexual HIV-concordant negative
* Cohabiting at least 3 months
* Both partners at least 18 years of age (women aged 18-45, men aged 18-65)
* Not on antiretroviral therapy including Post Exposure Prophylaxis (PEP) or Pre Exposure Prophylaxis (PrEP)
* Interested in participating
* Able and willing to provide informed consent (literacy is not required)
* Willing to complete interviewer-administered questionnaires on risk factors
* Available for follow-up for the duration of the study
* Willing and able to be contacted via phone or home visit
* Able and willing to provide adequate locator/contact information for retention purposes, and willing to be contacted by the study staff

Exclusion Criteria:

* Presence of any condition that, in the opinion of the investigator or designee, would preclude provision of informed consent, or otherwise interfere with achieving the study objectives
* Either partner HIV-positive or with indeterminate HIV rapid test results
* Attendance to a clinic involved in the opposite arm of the study (i.e., test with partner at a clinic indicated as SOV but attends a clinic indicated as GHPP or vice versa)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3450 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
HIV Incidence Rate | Duration of Study (Up to six months)
  The number of new laboratory confirmed HIV diagnosis.
Syphilis Incidence Rate | Duration of Study (Up to six months)
  The number of new laboratory confirmed syphilis diagnosis.
Vaginal Trichomoniasis Incidence Rate | Duration of Study (Up to six months)
  The number of new laboratory confirmed vaginal trichomoniasis diagnosis.
Number of Self-Reported Sexually Transmitted Infections (STIs) | Duration of Study (Up to six months)
  The number of self-reported STIs via questionnaire.
Number of Reports of Sex without a Condom with Outside Partners | Duration of Study (Up to six months)
  The number of reports of sex without using a condom reported via a study specific questionnaire.
Number of Reported Outside Partners | Duration of Study (Up to six months)
  The self-reported number of sexual partners outside of marriage.
Knowledge and use of hygiene and sanitation measures | Duration of Study (Up to six months)
  Number of participants who show increased knowledge of hygiene and sanitation measures via a study specific questionnaire.
Knowledge of hypertension and diabetes screening and management | Duration of Study (Up to six months)
  Number of participants who show increased knowledge of hypertension and diabetes screening and management via a study specific questionnaire.
Number of self-reports of accessing couples' testing (CVCT) with outside partners | Duration of Study (Up to six months)
  Number of participants who report accessing CVCT services with their outside partners reported via a study specific questionnaire.

SECONDARY OUTCOMES:
Perceived Efficacy of Chlorine Use | Duration of Study (Up to six months)
  The number of participants who report a perceived effect of chlorine use via a study specific questionnaire.
Perceived Efficacy of Handwashing | Duration of Study (Up to six months)
  The number of participants who report a perceived effect of handwashing via a study specific questionnaire.
Perceived Efficacy of Deworming | Duration of Study (Up to six months)
  The number of participants who report a perceived effect of deworming via a study specific questionnaire.
Perceived Efficacy of Management of Diabetes | Duration of Study (Up to six months)
  The number of participants who report a perceived effect of management of diabetes via a study specific questionnaire.
Perceived Efficacy of Management of Hypertension | Duration of Study (Up to six months)
  The number of participants who report a perceived effect of management of hypertension via a study specific questionnaire.
Change in Communication between Husband and Wife | Duration of Study (Up to six months)
  Change in communication between husband and wife dyads regarding exposure to HIV through extramarital sexual behaviors will be measured using a study specific questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Allen, MD, MPH, Principal Investigator — Emory University
Locations (2):
- Zambia (2):
  - Ndola Research Site, Ndola, Copperbelt
  - Lusaka Research Site, Lusaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharkey T, Parker R, Wall KM, Malama K, Pappas-DeLuca K, Tichacek A, Peeling R, Kilembe W, Inambao M, Allen S. Use of "Strengthening Our Vows" Video Intervention to Encourage Negotiated Explicit Sexual Agreements in Zambian Heterosexual HIV Seroconcordant-Negative Couples. Arch Sex Behav. 2023 Aug;52(6):2649-2667. doi: 10.1007/s10508-023-02590-x. Epub 2023 Apr 6. PMID 37024634